CLINICAL TRIAL: NCT03924323
Title: A Randomized, Multicenter, Double-Blind, Flexibly-dosed, Efficacy and Safety Study of Escitalopram in the Treatment of Children and Adolescents With Generalized Anxiety Disorder
Brief Title: A Study of Escitalopram in the Treatment of Children and Adolescents With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCT-MD-60
Record Dates: First submitted 2019-04-19; First posted 2019-04-23 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Anxiety Disorders,Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Escitalopram 10 mg/day (Experimental): Oral administration with the possibility of dose escalation to 20 mg/day at the investigator's discretion
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Matching oral administration of placebo once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Escitalopram — 8-weeks of treatment followed by 1-week taper down period
  Arms: Escitalopram 10 mg/day
Other: Placebo — Matching oral administration of inactive substance once daily
  Arms: Placebo

SUMMARY:
This is a study in minors (7 to 17 years old) diagnosed with generalized anxiety disorder (GAD) and evaluated using standard questionnaires as having at least moderate severity of GAD. Participating minors will be assigned to receive either the study drug escitalopram or a pill without any drug in it called a placebo. The purpose of this research is to study the safety and effectiveness of escitalopram in minors with GAD.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent/legal representative must give written informed consent, including privacy authorization, prior to study participation. The subject will complete an informed assent prior to study participation.
* Subject meets DSM-5 criteria for a primary diagnosis of GAD at screening established by a comprehensive psychiatric evaluation and confirmed/supported using the Mini-International Neuropsychiatric Interview for children and adolescents (MINI Kid).
* Male subjects who are sexually active with a partner of childbearing potential must use, with their partner, a condom plus an approved method of highly effective contraception from the time of informed consent until 14 days after the last dose of study drug.
* Female subjects who are sexually active and are of childbearing potential must use, with their partner, an approved method of highly effective contraception from the time of informed consent until 14 days after the last dose of study drug.
* Female subjects who are not of childbearing potential do not need to use any methods of contraception. This includes preadolescent and adolescent females who have not reached menarche. - Subject must have venous access enough to allow blood sampling and be compliant with blood draws as per the protocol.

Exclusion Criteria:

* Current diagnosis of MDD, attention-deficit/hyperactivity disorder, or lifetime diagnosis of bipolar disorder, psychotic depression, schizophrenia or other psychotic disorder, feeding and/or eating disorder, obsessive-compulsive disorder, conduct disorder, oppositional defiant disorder, post-traumatic stress disorder, panic disorder, or pervasive development disorder.
* Suspected or previously diagnosed intellectual disability disorder.
* One or more first-degree relatives with diagnosed bipolar I disorder.
* History of seizure disorder (other than febrile seizures).
* History of electroconvulsive therapy at any time during the subject's lifetime.
* Known hypersensitivity to escitalopram (escitalopram oxalate) or citalopram or any of the inactive ingredients or had frequent or severe allergic reactions to multiple medications.
* Taking any medications that are contraindicated to escitalopram (escitalopram oxalate).
* Inability to speak, read, or understand English well enough to complete the assessments.
* No active suicidal ideation or lifetime history of suicidal behavior as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 273 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (39):
- United States (39):
  - Harmonex /ID# 233342, Dothan, Alabama
  - Woodland International Research Group /ID# 233348, Little Rock, Arkansas
  - Woodland Research Northwest, LLC /ID# 233366, Rogers, Arkansas
  - ATP Clinical Research, Inc /ID# 233362, Costa Mesa, California
  - ProScience Research Group /ID# 233374, Culver City, California
  - Sun Valley Research Center /ID# 233343, Imperial, California
  - MCB Clinical Research Centers /ID# 233372, Colorado Springs, Colorado
  - Emerson Clinical Research Inst /ID# 233371, Washington D.C., District of Columbia
  - Innovative Clinical Research /ID# 233365, Fort Lauderdale, Florida
  - Indago Research and Health Cen /ID# 233364, Hialeah, Florida
  - CNS Healthcare - Jacksonville /ID# 233352, Jacksonville, Florida
  - Accel Research Sites-Maitland Clinical Research Unit /ID# 233368, Maitland, Florida
  - Medical Research Group of Central Florida /ID# 233357, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc /ID# 233350, Orlando, Florida
  - APG Research, LLC /ID# 233337, Orlando, Florida
  - University of South Florida Rothman Center of Neuropsychiatry /ID# 233356, St. Petersburg, Florida
  - Capstone Clinical Research /ID# 233354, Libertyville, Illinois
  - Baber Research Group /ID# 233363, Naperville, Illinois
  - Psychiatric Associates /ID# 233360, Overland Park, Kansas
  - Alivation Research /ID# 233338, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine Inc /ID# 233355, Las Vegas, Nevada
  - Manhattan Behavioral Medicine PLLC /ID# 233351, New York, New York
  - Finger Lakes Clinical Research /ID# 233347, Rochester, New York
  - Quest Therapeutics of Avon Lake /ID# 233367, Avon Lake, Ohio
  - Neuro-Behavioral Clinical Research, Inc. /ID# 233375, Canton, Ohio
  - University of Cincinnati /ID# 233341, Cincinnati, Ohio
  - UH Cleveland Medical Center /ID# 233373, Cleveland, Ohio
  - Midwest Clinical Research Center /ID# 233346, Dayton, Ohio
  - CincyScience /ID# 233359, West Chester, Ohio
  - SP Research, PLLC /ID# 233340, Oklahoma City, Oklahoma
  - Central States Research /ID# 233339, Tulsa, Oklahoma
  - Coastal Carolina Research Center /ID# 233344, North Charleston, South Carolina
  - Houston Clinical Trials /ID# 233345, Bellaire, Texas
  - Relaro Medical Trials /ID# 233369, Dallas, Texas
  - AIM Trials /ID# 233361, Plano, Texas
  - Focus Center, PC /ID# 233349, Ogden, Utah
  - University of Virginia /ID# 233370, Charlottesville, Virginia
  - Northwest Clinical Research Center /ID# 233358, Bellevue, Washington
  - Core Clinical Research /ID# 233353, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Strawn JR, Moldauer L, Hahn RD, Wise A, Bertzos K, Eisenberg B, Greenberg E, Liu C, Gopalkrishnan M, McVoy M, Knutson JA. A Multicenter Double-Blind, Placebo-Controlled Trial of Escitalopram in Children and Adolescents with Generalized Anxiety Disorder. J Child Adolesc Psychopharmacol. 2023 Apr;33(3):91-100. doi: 10.1089/cap.2023.0004. PMID 37074330

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 273 participants are included in the Safety Population with 136 participants being randomized to the Placebo group and 137 participants randomized to the Escitalopram group
Period: Overall Study
Arm/Group | Placebo | Escitalopram 10 mg/Day
Started | 136 | 137
Completed | 117 | 123
Not Completed | 19 | 14

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of all subjects in the Randomized Population who took at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Escitalopram 10 mg/Day | Total
Number analyzed (Participants) | 136 | 137 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (2.6) | 12.7 (2.7) | 12.6 (2.6)
Age, Customized [Count of Participants; unit: Participants]
  7 Years to 11 Years | 45 | 44 | 89
  12 Years to 17 years | 91 | 93 | 184
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 94 | 187
  Male | 43 | 43 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 31 | 53
  Not Hispanic or Latino | 114 | 106 | 220
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 15 | 13 | 28
  White | 110 | 113 | 223
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Pediatric Anxiety Rating Scale (PARS) Severity Score
Description: The PARS is a clinician-rated instrument for assessing the severity of anxiety symptoms associated with common anxiety disorders including generalized anxiety disorder (GAD) in children. The PARS severity score for GAD will be assessed for all symptoms identified in the generalized anxiety section of the PARS symptom checklist derived by summing 5 of the 7 severity/impairment/interference items (2, 3, 5, 6, and 7) each item ranged from 0 (none) to 5 (extreme severity/impairment/interference). PARS severity scores for GAD ranged from 0 (none) to 25 (extreme severity), with a score of 15 indicating moderate illness severity.
Time Frame: Baseline to Week 8
Population: The modified Intent-to-treat (mITT) Population was defined as all subjects who were randomized and received at least 1 dose of study medication and had both baseline and at least 1 post-baseline primary efficacy measure (ie, PARS severity score).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Escitalopram 10 mg/Day
Number analyzed (Participants) | 117 | 124
score on a scale | -6.38 (0.494) | -7.81 (0.484)
Statistical Analysis 1: Comparison: Placebo vs Escitalopram 10 mg/Day; Test type: Superiority; p = 0.0281, mixed-effects model for repeated measure; least squares mean difference = -1.42, 95% CI 2-sided [-2.69 to -0.15]

2. Secondary Outcome: Response Rate on the PARS
Description: Response is defined as a 50% improvement on the PARS severity score for GAD
Time Frame: Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Escitalopram 10 mg/Day
Number analyzed (Participants) | 117 | 124
Participants | 39 | 49
Statistical Analysis 1: Comparison: Placebo vs Escitalopram 10 mg/Day; Test type: Superiority; p = 0.4521, generalized linear mixed model (GLMMIX); Odds Ratio (OR) = 1.253, 95% CI 2-sided [0.695 to 2.258]

3. Secondary Outcome: Remission Rate on the PARS
Description: Remission is defined as PARS severity score for GAD ≤8 (using 6 PARS items: 2, 3, 4, 5, 6, and 7)
Time Frame: Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Escitalopram 10 mg/Day
Number analyzed (Participants) | 117 | 124
Participants | 22 | 22
Statistical Analysis 1: Comparison: Escitalopram 10 mg/Day; Test type: Superiority; p = 0.6928, generalized linear mixed model (GLMMIX); Odds Ratio (OR) = 1.157, 95% CI 2-sided [0.560 to 2.387]

4. Secondary Outcome: Change on the Clinical Global Impression of Severity (CGI-S)
Description: Remission rate on CGI-S at acute treatment endpoint (Week 8). Remission rate is defined as the percentage of subjects having a CGI-S score ≤2 at endpoint. CGI-S is a seven point scale where 1=Normal and 7=Among the most extremely ill patients.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Escitalopram 10 mg/Day
Number analyzed (Participants) | 118 | 124
score on a scale | -1.2 (1.1) | -1.3 (1.0)

5. Secondary Outcome: Change on the Children's Global Assessment Scale (CGAS)
Description: Remission rate on the CGAS at acute treatment endpoint (Week 8). Functional remission is defined as CGAS >70. The CGAS used is a 100-point scale ranging from 1 to 100, with higher scores indicating better functioning.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Escitalopram 10 mg/Day
Number analyzed (Participants) | 118 | 124
score on a scale | 16.2 (12.9) | 18.1 (13.1)

ADVERSE EVENTS:
Time Frame: All AEs from the time the subject signed the ICF until 30 days after receiving the last dose of study drug were collected (Up to 10 weeks).
Groups:
- Escitalopram 10 mg/Day: Oral administration with the possibility of dose escalation to 20 mg/day at the investigator's discretion Escitalopram: 8-weeks of treatment followed by 1-week taper down period
- Placebo: Matching oral administration of placebo once daily Placebo: Matching oral administration of inactive substance once daily
Arm/Group | Escitalopram 10 mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/136
Serious Adverse Events (participants affected / at risk) | 2/137 | 1/136
Other Adverse Events (participants affected / at risk) | 44/137 | 27/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram 10 mg/Day (N=137) | Placebo (N=136)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 2 (2) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram 10 mg/Day (N=137) | Placebo (N=136)
NAUSEA (Gastrointestinal disorders) | 18 (19) | 7 (8)
FATIGUE (General disorders) | 7 (8) | 10 (10)
DECREASED APPETITE (Metabolism and nutrition disorders) | 10 (10) | 4 (4)
HEADACHE (Nervous system disorders) | 10 (13) | 10 (12)
SOMNOLENCE (Nervous system disorders) | 7 (7) | 2 (2)
INSOMNIA (Psychiatric disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT03924323/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03924323/SAP_001.pdf